# **Statistical Analysis Plan**

| Date: | 06-Mar-2024 |
|----------|-------------|
| Version: | v01 |
| Status: | final |
| Author: | |

Study Title: A phase 2 trial of EO2040, a miCrobiaL-derived

peptide therApeUtic vaccine, in combination with nivolumab, for treatment of patients with circulating tumor DNA-dEfined minimal residual disease of colorectal cancer stage II, III, or IV after completion

of curative therapy (the "CLAUDE" study).

Investigational Product: EO2040

Clinical Phase:

Enrolment of first patient 19-Jan-2023 (actual date)

Last Patient Last Visit 23-Jan-2024 (actual date)

Sponsor: Enterome

94/96 avenue Ledru-Rollin 75011

Paris, France

Project Manager (Sponsor):

Data Management and Biostatistics (CRO):

Project Manager :

Lead Statistician :

Supervisor Biostatistics

Enterome: EOCRC1-22

(EN05) 

# **Signatures**



Version/Status/Date: v01/final/06-Mar-2024

Enterome: EOCRC1-22

(EN05) 

# **Table of Contents**

| Si | ignatur | es | | | 2 |
|---|---|---|---|---|---|
| Tá | able of | Contents | | | 3 |
| 1 | Do | cument History | | | 4 |
| 2 | List | t of Abbreviations | | | 4 |
| 3 | Ger | neral | | | 5 |
| | 3.1 | Analyses Planned and Already Performed | 5 | | |
| | 3.2 | SOPs to be Followed | 5 | | |
| 4 | Ove | erview of the Protocol | | | 5 |
| | 4.1 | Study Objectives | 5 | | |
| | 4.1 | - // | | 5 | |
| | 4.1<br>4.1 | | | 5<br>6 | |
| | 4.1 | .3 Exploratory Objectives Study Endpoints | 6 | O | |
| | 4.2 | • | 0 | 6 | |
| | 4.2 | · · | | 7 | |
| | 4.2 | .3 Exploratory Endpoint | | 7 | |
| | 4.3 | Study Design | 8 | | |
| | 4.4 | Sample Size | 10 | | |
| | 4.5 | Study Flow Chart | 10 | | |
| 5 | Gei | neral Aspects of the Statistical Analysis | | 1 | 1 |
| | 5.1 | Analysis Sets | 11 | | |
| | 5.2 | Protocol Devations | 11 | | |
| | 5.3 | Intercurrent Events | 11 | | |
| | 5.4 | Changes or Deviations from Planned Analyses | 11 | | |
| 6 | Def | initions for Statistical Analysis | | 1 | 1 |
| | 6.1 | Baseline and Change from Baseline | 11 | | |
| | 6.2 | Study Day | 11 | | |
| | 6.3 | Duration | 12 | | |
| | 6.4 | Visit windows and Analysis Visits | 12 | | |
| 7 | Sta | tistical Analysis Specification | | 1 | 2 |
| | 7.1 | Specifications Related to Whole Analysis | 12 | | |
| | 7.1 | | | 12 | |
| | 7.1 | 3.5 | | 12 | |
| 8 | | tware and Statistical Programming | | | |
| 9 | | erences | | | |
| 10 | | anges to Final Version of the SAP | | | |
| 11 | | t of Tables, Figures and Listings | | 1 | 4 |
| | 11.1 | Table of Contents for End-of-Text Tables and Figures | | | |
| | 11.2 | Table of Contents of Individual Patient Data Listings (Appendix 16.2 of the CSR) | | | |
| | 11.3 | Grading of safety laboratory parameters analogous to NCLCTCAF v5.0 | 15 | | |


#### 1 DOCUMENT HISTORY

| Version | Date | Author / editor of new version | Main changes / comments |
|---|---|---|---|
| v01 | 06-Mar-2024 | | First version |

#### 2 LIST OF ABBREVIATIONS

| Λh | araviation | OVI |
|-----|------------|------|
| ~~~ | breviation | Text |

AE Adverse Events
APS All-Patient Set

ATC Anatomical Therapeutic Chemical

BIRC5 Baculoviral Inhibitor of Apoptosis Repeat-containing5

CRC Colorectal cancer
CRF Case Report Form
CSR Clinical Study Report

ctDNA Circulating tumor deoxyribonucleic acid

DFS Disease-free survival
DNA Deoxyribonucleic acid
eCRF Electronic Case Report

eCRF Electronic Case Report Form ELISpot Enzyme-linked Immunospot

FAS Full Analysis Set FOXM1 forkheadboxM1

ICH International Council for Harmonization

IFN-γ Interferon-gamma
IHC Immunohistochemistry

MDSC Myeloid-derived suppressor cells

MedDRA Medical Dictionary for Regulatory Activities

MRD Minimal residual disease

NCI-CTCAE

National Cancer Institute-Common Terminology Criteria for

ΑE

OS Overall Survival

PD-L1 Programmed Death-Ligand 1

PPS Per-Protocol Set
PT Preferred Term
QC Quality control

SAE Serious Adverse Event

SOC Standard of Care, System Organ Class

SOP Standard Operating Procedure

SS Safety Set

TAA Tumor associated antigens

TCR T cell Receptor

TEAE Treatment-Emergent Adverse Events

UCP2 Universal Cancer Peptide 2

WHODD World Health Organization Drug Dictionary

based on

#### 3 GENERAL

This statistical analysis plan reflects study protocol EOCRC1-22 dated 04-JUL-2022. It follows the principles of the Guidelines International Council for Harmonization (ICH) Topic E3 and ICH Topic E9. It gives all details for the final statistical analysis of this study.

### 3.1 Analyses Planned and Already Performed

No formal analysis of the data will be performed as the study is planned to be terminated with just one treated patient, only patient data listings will be produced.

#### 3.2 SOPs to be Followed

The analysis will be carried out according to Metronomia Standard Operation Procedures (SOPs).

The report will be written according to the ICH E3 and other applicable ICH guidelines.

### 4 OVERVIEW OF THE PROTOCOL

## 4.1 Study Objectives

#### 4.1.1 Primary Objective

• The primary objective of this trial is to assess the 6-month circulating tumor deoxyribonucleic acid (ctDNA) clearance rate at therapy with EO2040 in combination with nivolumab, in patients with ctDNA-defined minimal residual disease (MRD) of stage II-IV colorectal cancer after completion of curative therapy.

and in sequence, provided the first objective has a positive outcome per protocol Section 9:

- The primary objective is, to assess the 6-month ctDNA clearance rate at therapy with EO2040 monotherapy, in patients with ctDNA-defined MRD of stage II-IV colorectal cancer after completion of curative therapy.
  - In case the first objective does not have a positive outcome per protocol Section
     9, a protocol amendment to adjust the second part of the primary objective to utilize an alternative therapeutic vaccine than EO2040 will be considered.

ctDNA clearance is utilized as a surrogate endpoint for eventual cure, and thereby prolongation of disease-free survival (DFS) for patients achieving clearance.

Note, clearance of ctDNA is characterized by the disappearance of all somatic mutations identified in the blood, as well as no appearance of any additional new somatic mutations, and radiographic investigation(s) showing no evidence of colorectal cancer (see protocol Section 7.8).

#### 4.1.2 Secondary Objectives

To assess the following items at therapy with EO2040 in combination with nivolumab, and when applicable EO2040 monotherapy, in patients with ctDNA-defined MRD of stage II-IV colorectal cancer after completion of curative therapy:

- Safety and tolerability of study treatments,
- The 3-month ctDNA clearance rate,


- Progression of colorectal cancer and death as DFS,
- Overall Survival (OS),
- Survival at 36 months after start of study therapy, and
- Induction/expansion of T cells specific for EO2040, the components of EO2040, and the targeted nominal tumor associated antigens (TAAs) (Baculoviral Inhibitor of Apoptosis Repeat-containing5 [BIRC5] and forkheadboxM1 [FOXM1]).

#### 4.1.3 Exploratory Objectives



### 4.2 Study Endpoints

#### 4.2.1 Primary Endpoint

 The primary endpoint is response to treatment at 6 months (see protocol Section 3.1.1), which is defined as having clearance of ctDNA, AND not having any radiographic evidence of recurrence at 6 months (see also protocol Section 7.8 for rules of assessment of an individual patient best overall response).

Clearance of ctDNA will be characterized by the disappearance of all somatic mutations

Enterome: EOCRC1-22 (EN05) 

identified in the blood, as well as no appearance of any additional new somatic mutations.

## 4.2.2 Secondary Endpoint

- The safety and tolerability of study treatments will be determined by a descriptive medical assessment of the combined profile of incidences of adverse events (AEs), treatment-emergent AEs (TEAEs), serious AEs (SAEs), deaths, reasons for treatment discontinuation/delays, and laboratory abnormalities using the NCI-CTCAE v5.0 grading system (see Section 11.3 below and Section 7.7 in protocol).
- Response to therapy at 3 months, defined as clearance of ctDNA, AND no radiographic evidence of recurrence (determination method will be the same as for the primary endpoint; see protocol Section 3.2.1).
- DFS defined as the time from start of study treatment to the date of first documented CRC recurrence or death due to any cause, whichever occurs first. Patients alive without recurrence will be censored at the date of last follow-up time. Recurrence is defined by the appearance of one or more new CRC lesions on imaging and/or other clinical evaluation such as endoscopy.
- OS, measured as the time from start of study treatment until death from any cause. Patients alive will be censored at the last time documented to be alive.
- Survival at 36 months after start of study treatment, estimated via Kaplan-Meier estimates.

Immunogenicity and cross reactivity: immunogenicity determined as expansion of

| | | | Γ cells<br>patien | comparing | samples | versus | on | treatment | in | ar |
|---|---|---|---|---|---|---|---|---|---|---|
| | ITATVIC | addi | patien | | | | | | | |
| Ex | plorate | ory | Endpo | int | | | | | | |

4.2.3

**Statistical Analysis Plan** 

Version/Status/Date: v01/final/06-Mar-2024

Enterome: EOCRC1-22 (EN05) 

| • | Correlations between immunogenicity |
|---|---|
| | of EO2317, EO2318, and UCP2 and clinical efficacy (per primary and secondary efficacy endpoints) and safety (TEAEs of defined specificities and grades) outcome parameters. Cross reactivities shown for the TAAs BIRC5/survivin, and FOXM1 will also be explored in the same way. |

#### 4.3 **Study Design**

The trial is a multi-center, open-label, non-comparative, two sequential cohort, phase 2 trial, to investigate as the first cohort efficacy of the microbiome-derived therapeutic vaccine EO2040 in combination with nivolumab in patients with stage II-IV colorectal cancer with ctDNA defined MRD after completion of curative therapy. Assuming a positive outcome of the first cohort, a second cohort assessing efficacy of EO2040 monotherapy, with the option of addition of nivolumab after 3 months in case of no ctDNA clearance, is planned.

The study is assumed to recruit a total of 17 patients in Cohort 1, and if cohort 1 has a positive outcome (see protocol Section 9), a total of 17 patients will also be recruited to Cohort 2A.

Schematic overview of the trial design, and an overview of the treatment schedule are illustrated in figures below.

#### Trial design overview:



Treatment schedule, scan and ctDNA assessments, and blood sampling for immune testing and serum collection:

Enterome: EOCRC1-22 (EN05)


#### 4.4 Sample Size

| Considering | prior a | attempts | in similar | situations, | the tri | al will | include | 17 | patients | per | cohort. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| The primary | object | ive of the | trial is to | determine | the ct[ | DNA cl | learance | rat | e at 6 m | onth | s (R6). |

| 1 |
|---|

#### **Study Flow Chart** 4.5

Refer the latest study protocol.

#### 5 GENERAL ASPECTS OF THE STATISTICAL ANALYSIS

### 5.1 Analysis Sets

The **All-Patient (AP) set** will consist of any patient who signed informed consent including screen-failures.

The **Full Analysis Set (FAS)** will consist of patients who received at least one dose of EO2040 and for whom no important protocol deviations occurred that would compromise the evaluation of efficacy.

The **Safety Set (SS)** will consist of patients who received at least one dose of study treatment.

#### 5.2 Protocol Devations

All protocol deviations regardless of their source will be listed for each patient together with the categorization into major or minor.

#### 5.3 Intercurrent Events

Not Applicable.

## 5.4 Changes or Deviations from Planned Analyses

Since the study is planned to be terminated with just one treated patient, no formal analysis of the data will be performed.

#### 6 DEFINITIONS FOR STATISTICAL ANALYSIS

#### 6.1 Baseline and Change from Baseline

Baseline is defined as the last non-missing value prior to first administration of study treatment.

Absolute Change from Baseline at a visit/timepoint will be calculated as follows:

Result at visit/timepoint – Baseline result;

For assessments taken before and after first administration of study treatment, baseline assessments will be flagged separately in the listings. Similarly, change from baseline values will be displayed alongside observed results in the respective listings.

#### 6.2 Study Day

The reference day (Day 1) for study day calculations is the date of the first administration (V1) of study treatment. The study day will be calculated as follows:

- Assessment/Visit Date Date of first administration study treatment + 1; for assessments on or after the date of first administration of study treatment
- Assessment/Visit Date Date of first administration study treatment; for assessments before the date of first administration of study treatment


There is no Study Day 0.

Study day will be displayed alongside visit/event dates in the relevant listings.

#### 6.3 Duration

Duration of an event will be calculated as follows:

Duration (days) = (End date of event - Start date of event) +1;

In case of partial start/end dates, duration will be calculated assuming the 15<sup>th</sup> of the respective months if case of missing day. Duration will not be calculated if months and day are not given.

All listings displaying event data like AE, medication, etc., will include duration of the events alongside the end dates.

#### 6.4 Visit windows and Analysis Visits

Data collected by visit will be displayed for the visit it was collected, irrespective of the actual date of the assessment.

The following tables shows the visit labels to be used in patient data listings:



#### 7 STATISTICAL ANALYSIS SPECIFICATION

## 7.1 Specifications Related to Whole Analysis

#### **7.1.1 Tables**

No tables will be produced.

#### 7.1.2 Data Listings

All CRF data will be listed as documented. For screen failures only demographic data and screen failure details will be listed. Relevant generated variables from section 6 will be listed


next to the original data items as well.

In all listings, the cohort labels will be displayed as given below:

- Cohort 1
- Cohort 2A
- Cohort 2B

In listings with screen failure data, screen failures will have cohort label as "Not Applicable" and will be sorted at last.

The listings will be sorted by cohort, patient identifier, visit and date (if applicable).

#### Medical history, Procedures and Adverse event:

All medical history, concomitant illness, procedures and adverse events will be coded using MedDRA version mentioned in the latest data management plan and system organ class (SOC), preferred term (PT) of the events will be presented in the listing.

#### Medication:

All medication will be coded using World Health Organization Drug Dictionary (WHODD) version mentioned in the latest data management plan and Anatomical Therapeutic Chemical (ATC) level 2 term, PT of the medications will be presented in the listing.

#### 8 SOFTWARE AND STATISTICAL PROGRAMMING

The statistical analysis will be performed using the SAS® statistical software package in Version 9.4.

SAS programming will be performed according to Metronomia standards as defined in BM-08-SOP "Statistical Analysis and Programming" and related work instructions. Special attention will be paid to planning and performance of quality control measures as documented in the QC plan for the analysis of this study (see also BM-08-WIN03 "How to Plan and Document QC for Statistical Analysis").

#### 9 REFERENCES

Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, Published: November 27, 2017. U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES, National Institutes of Health National Cancer Institute, https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/ctcae\_v5\_quick\_r eference\_5x7.pdf. Accessed February 2, 2024.

ICH Topic E9: Statistical Principles for Clinical Trials, 5 February 1998, adopted by CPMP, March 1998, issued as CPMP/ICH/363/96ICH

ICH E9 (R1): Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials, 20 November 2019, adopted by CHMP, 30 January 2020, issued as EMA/CHMP/ICH/436221/2017

SAS 9.4 https://support.sas.com/documentation/94/index.html. Copyright © SAS Institute Inc., SAS Campus Drive, Cary, North Carolina 27513, USA. All rights reserved.

**Statistical Analysis Plan** 

Version/Status/Date: v01/final/06-Mar-2024

Enterome: EOCRC1-22 (EN05)


#### **CHANGES TO FINAL VERSION OF THE SAP** 10

Not Applicable.

#### **LIST OF TABLES, FIGURES AND LISTINGS** 11

#### 11.1 **Table of Contents for End-of-Text Tables and Figures**

No tables and figures will be produced.

#### 11.2 Table of Contents of Individual Patient Data Listings (Appendix 16.2 of the CSR)



Enterome: EOCRC1-22

(EN05)




Grading of safety laboratory parameters analogous to NCI CTCAE v5.0 11.3

Enterome: EOCRC1-22

(EN05)


